CLINICAL TRIAL: NCT03617237
Title: Registry Study to Evaluate the Clinical Outcome of Cancer Patients and Benign Diseases Treated with Radiation At the University of Texas Southwestern Medical Center
Brief Title: Registry Study to Evaluate the Clinical Outcome of Cancer Patients and Benign Diseases Treated with Radiation
Status: Recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, David Sher, Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU 052012-019
Record Dates: First submitted 2018-05-14; First posted 2018-08-06 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Retrospective Populations — All patients who are currently treated by any physician at the University of Texas Southwestern campus Aston Clinic, Seay Clinic, PHHS Clinic, Moncrief Radiation Oncology, St. Paul West Campus Radiation Oncology, East Radiation Oncology Clinic will be included in the registry. The data from the charts will be entered into a password protected excel spreadsheet. The charts will be identified by name, medical record number, date of birth, and social security number.
  1. The research involves no more than minimal risk to the subjects.
  2. The waiver will not adversely affect the rights and welfare of the subjects.
  3. The research could not practicably be carried out without the waiver.
  4. Whenever appropriate, the subjects will be provided with additional pertinent information after participation.

SUMMARY:
Registry database repository for determining clinical outcomes primarily of patients who have received or have been evaluated for radiation treatment in either the definitive or palliative setting for both malignant and benign etiologies.

To compare the outcomes with National Cancer Data Base (NCDB) of the American College of Surgeon(ACS).

DETAILED DESCRIPTION:
Investigator will retrospectively collect and evaluate information from patients with cancer or benign etiologies to improve future clinical outcomes and help identify prospective outcomes study questions. This information will include patients' name, medical record number, medical history, diagnosis, treatment, laboratory test results, diagnostic test results, pathology reports, therapeutic and nontherapeutic results, surgical results, radiology results, radiation therapy details (dose, techniques, toxicity), concurrent use of chemotherapy/systemic therapy, quality of life outcomes,cachexia status, and primarily last follow-up data. All information will be collected after their standard of care visits.

ELIGIBILITY:
Inclusion Criteria:

Any patient who received or was potentially evaluated for radiotherapy since 2000 for benign or malignant etiologies in the definitive or palliative setting.

Patients with comparatively similar diagnosis and disease status at UTSW, but electing not to undergo radiation therapy, treated with surgical or systemic therapy, or best supportive care, being followed by an oncology specialist at UT Southwestern Medical Center will also be eligible for evaluation. -

Exclusion Criteria:

None

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Risk will be minimized by protecting patient data through the use of deidentification of patient identifiers and password protected data collection. The information will be given only to faculty members and statisticians involved in the research project. The information will include the parameters attached in the spreadsheet supplied with the IRB submission. The data will be disclosed only for analytical purposes.Confidentiality will be maintained by adhering to HIPAA guidelines. Only the PI and other study team members will have access to that data.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2012-07-03 (Actual); Primary Completion 2030-07-10 (Estimated); Study Completion 2032-04-18 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Analysis | 10 years
  The quality of life questionnaire will be used as a standardized instrument to measure the health outcome.Its provides a simple descriptive profile and a single index value for health status. The US version of the EQ-5D will be used, to enable mapping of general HR-QOL scores from EQ-5D scores into health state utility scores (ranging from 0 to 100) for the US population.Analyses will be performed for all subjects having received treatment for benign and cancer tumors. Information gained from this could lead to improved medical care for them. By performing comparative study for subgroups of patients with similar diseases but not treated with radiation therapy, potential benefits and risks of radiation therapy may be better delineated.

CONTACTS AND LOCATIONS:
Overall Officials: David J Sher, MD, MPH, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Centre, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided